CLINICAL TRIAL: NCT04561076
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Phase I Clinical Study to Evaluate Safety and Pharmacokinetics of HLX70 in Healthy Adult Volunteers
Brief Title: Evaluate Safety and Pharmacokinetics of HLX70 in Healthy Adult Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor strategy
Sponsor: Hengenix Biotech Inc (Industry)
Collaborators: Sanyou Biopharmaceuticals(Shanghai)Co., Ltd (Unknown); Shanghai ZJ Bio-Tech Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: HLX70-001US-255086
Record Dates: First submitted 2020-09-07; First posted 2020-09-23 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind, Placebo-Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence 1 (Experimental): Random allocation to HLX70 3 mg/kg (IV, single dose), or placebo (IV, single dose) of which 2 receive intravenous injections of placebo and 6 receive intravenous injections of the HLX70.
  Interventions: Drug: HLX70; Other: Placebo
- Sequence 2 (Experimental): Random allocation to HLX70 10 mg/kg (IV, single dose), or placebo (IV, single dose) of which 2 receive intravenous injections of placebo and 6 receive intravenous injections of the HLX70.
  Interventions: Drug: HLX70; Other: Placebo
- Sequence 3 (Experimental): Random allocation to HLX70 30 mg/kg (IV, single dose), or placebo (IV, single dose) of which 2 receive intravenous injections of placebo and 6 receive intravenous injections of the HLX70.
  Interventions: Drug: HLX70; Other: Placebo

INTERVENTIONS:
Drug: HLX70 — Single-dose, intravenous infusion
  Other Names: Anti-spike protein-1 monoclonal antibody (mAb)
Other: Placebo — Single-dose, intravenous infusion

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Phase I Clinical Study to Evaluate Safety and Pharmacokinetics of HLX70 in Healthy Adult Volunteers

DETAILED DESCRIPTION:
A randomized, double-blind, single-dose by intravenous administration, placebo-controlled, dose escalation, first-in-human study is proposed to evaluate the safety, PK, and immunogenicity of HLX70 in healthy subjects. The investigators plan to enroll 8 subjects in each of the 3 dose cohorts at 3 mg/kg, 10 mg/kg, and 30 mg/kg, of which 2 receive intravenous injections of placebo and 6 receive intravenous injections of the investigational product (IP). A total of 24 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with voluntary signing of the informed consent form (ICF);
2. Healthy males or females aged ≥ 18 and ≤ 60 years at the time of signing the ICF;
3. Subjects with body weight ≥ 50 kg and body mass index (BMI) must be higher than 18.5 kg/m2 and lower than 30 kg/m2 at screening visit;
4. Subjects who are determined to be in good health according to medical history, normal (site normal ranges to be followed) or abnormal but clinically insignificant physical examination, vital signs, ECG, laboratory test results (including hematology, serum chemistry, coagulation function, urinalysis, etc.), and investigator's clinical judgment (CTCAE grade 1 of triglycerides and uric acid is permitted). One re-test allowed per investigator discretion to confirm result.
5. Subject who agrees that he/she, and his/her spouse or partner, will use reliable contraception (see appendix 1) for 9 months after administration.

Exclusion Criteria:

1. Subjects with the lab-confirmed medical history of COVID-19, including nucleic acid (PCR testing of nasopharyngeal samples) tested positive or antibody IgG/IgM tested positive.
2. Subjects with the novel onset of pyrexia/cough/shortness of breath/diarrhea or history of contact with confirmed COVID-19 individuals (positive for SARS-CoV-2 nucleic acid) within the 14 days before randomization.
3. Subjects who are known to have chronic obstructive pulmonary disease (COPD), cirrhosis of liver, cardiac failure or any condition that requires active medical intervention or monitoring to avert serious danger to the participant's health or well-being.
4. Subjects with pneumonia or tuberculosis (TB) suggested by chest X-Ray.
5. Subjects with previous exposure to a mAb or any other biological agents in 6 months before screening.
6. Subjects with previous exposure to vaccines in 3 months before screening, or who plans to receive vaccination during the study period or in 3 months after the study.
7. Subjects with previous participation in clinical trials receiving investigational drug/comparator within the longer of 30 days or 5 half-lives before screening.
8. Subjects who are known to have a history of allergy to any mAb, biological product, protein product, or the ingredient of the IP.
9. Subjects with positive test result(s) for hepatitis B virus (positive for HBsAg or positive for HBcAb and HBV-DNA), hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV) antibodies, or treponema pallidum.
10. Subjects who are known to have a history of psychotropic drug abuse, alcoholism, or drug addiction within the last year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-09 (Estimated); Primary Completion 2021-09-06 (Estimated); Study Completion 2021-09-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events, serious adverse event and infusion-related reactions as assessed by CTCAE v5.0 | up to 92 days
Safety evaluation- proportion of subjects undergoing DLT events | Days 1 to 7
  The proportion of subjects undergoing DLT events

SECONDARY OUTCOMES:
PK parameters-Areas under the concentration-time curves | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
PK parameters-Maximum measured concentration | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
PK parameters-Time from dosing to maximum measured concentration | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
PK parameters-Terminal phase elimination rate constant | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
PK parameters-Terminal phase elimination half life | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
PK parameters-Clearance | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
PK parameters-Volume of distribution during terminal phase and at steady state | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
PK parameters-Mean residence time | pre-infusion (pre-dose), immediately post-infusion, 3 hours, 6 hours and 10 hours post-infusion, Days 2, 3, 5, 8, 11, 15, 22, 29, 43, 57, 71 and 92.
Anti-drug antibody | pre-infusion and Days 15, day 29, day 57, and day 92
  The number of presence subjects that develop of anti-durg antibody (immunogenicity)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Yoon, MD, Principal Investigator — California Clinical Trials Medical Group (CCTMG) managed by Parexel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343